CLINICAL TRIAL: NCT06421259
Title: To Switch or Not to Switch to CAB/RPV in PLWH With Past HBV Infection? Risk of HBV Reactivation? A Need for New HBV Markers?
Brief Title: Descriptive Analysis of Changes in Hepatitis B Markers in People Living With HIV on Injectable Therapy.
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Infectio01
Record Dates: First submitted 2024-05-13; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-03

CONDITIONS: Hiv Infection; Hepatitis B
MeSH Terms: conditions — HIV Infections; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV infected patients under injectable ART: HIV infected patients under injectable ART

SUMMARY:
In order to assess the risk of hepatitis B reactivation in people living with HIV and undergoing injection therapy, we propose to carry out a descriptive analysis of the evolution of hepatitis B markers in this population.

ELIGIBILITY:
Inclusion Criteria:

-HIV infected patients under injectable ART

Exclusion Criteria:

-Active HBV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients attending care in the infectiious disease department of the Universitary Hospital of Nice
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Risk of HBV reactivation under injectable HIV ART | From start of injectable HIV treatment to hepatitis B reactivation, assessed up to 24 months
  HBV serology, DNA HBV levels

CONTACTS AND LOCATIONS:
Overall Officials: Alissa NAQVI, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU NiICE, Nice, Alpes Maritimes, France